CLINICAL TRIAL: NCT00691457
Title: Comparison of 3 Novel Contact Lens Solutions on the Basal Lamina
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMA-08-09
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2009-06

CONDITIONS: Contact Lens Solution
Keywords: Contact lens; solution; confocal microscope

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Opti-Free contact lens solution
  Interventions: Device: Opti-Free contact lens solution
- 2 (Active Comparator): ReNu Multiplus contact lens solution
  Interventions: Device: ReNu Multiplus contact lens solution
- 3 (Active Comparator): Clear Care contact lens solution
  Interventions: Device: Clear Care contact lens solution

INTERVENTIONS:
Device: Opti-Free contact lens solution — Solution
  Arms: 1
Device: ReNu Multiplus contact lens solution — Solution
  Arms: 2
Device: Clear Care contact lens solution — Solution
  Arms: 3

SUMMARY:
Three arm study comparing three novel contact lens solutions.

ELIGIBILITY:
Inclusion:

* Stable distance contact lens prescription between -0.50 D and 9.00 D and astigmatism less than or equal to -1.00 D cylindrical (cyl).
* Stable correction is defined as longer than six months.
* Worn a single brand of disposable silicone hydrogel contact lenses successfully (i.e., without complications or discomfort) for a minimum of six months

Exclusion:

* Known sensitivity to the contact lens disinfecting solutions or fluorescein dye.
* Any systemic or ocular disease that could affect contact lens wear.
* Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in corneal fluorescein staining as evaluated at Day 30 | 30 Days

SECONDARY OUTCOMES:
Confocal evaluation variables as measured at Days 0, 14, and 30 | Day 0, 14, 30

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Beach, VA, Virginia Beach, Virginia, United States